CLINICAL TRIAL: NCT04102280
Title: Comparative Clinical Performance of Dialyzers Applied During High Volume Online Haemodiafiltration - comPERFORM Study (Comparative PERFORMance)
Brief Title: Comparative Clinical Performance of Dialyzers Applied During High Volume Online Haemodiafiltration
Acronym: comPERFORMStud
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Institut Dr. Schauerte (IDS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HD-FX-07-D
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Renal Failure; End Stage Renal Disease
Keywords: Hemodialysis; Hemodiafiltration; Renal replacement therapy
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Kidneys, Artificial

STUDY DESIGN:
Intervention Model Description: prospective, open, controlled, cross-over (with randomized treatment sequences), interventional, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodiafiltration HDF (Other): Three consecutive treatment weeks and one follow-up week per patient. Each treatment week includes three hemodiafiltration HDF sessions and is assigned to one type of dialyzer: FX P600 Fresenius Medical Care, comparator Xevonta Hi 15 (B. Braun) and comparator Elisio 150H (Nipro)
  Interventions: Device: Dialyser

INTERVENTIONS:
Device: Dialyser — Three consecutive treatment weeks and one follow-up week per patient. Each treatment week includes three hemodiafiltration HDF sessions and is assigned to one type of dialyzer: FX P600 Fresenius Medical Care, comparator Xevonta Hi 15 (B. Braun) and comparator Elisio 150H (Nipro)

SUMMARY:
The clinical investigation will be performed to generate clinical data on clearances and removal rates for ß2-microglobulin and other uremic toxins and on clinical adverse events of the modified polysulfone membrane to fulfil obligations to follow the FX P600 dialyzer in the market.

DETAILED DESCRIPTION:
The primary objective of this study is to test whether the FX P600 is non-inferior to the Xevonta Hi 15 dialyzer and the Elisio 150H dialyzer in removing β2-microglobulin related to the albumin removal into the dialysate during high volume online hemodiafiltration.

The secondary objective of this study is to compare the FX P600 dialyzer with the comparator dialyzers with regard to their efficacies in removing other performance variables (see below). Furthermore, the safety of the FX P600 will be investigated by collecting and analyzing clinical adverse events.

ELIGIBILITY:
Inclusion Criteria:

General:

* Informed consent signed and dated by study patient and investigator/authorized physician
* Minimum age of 18 years
* Legally competent and able to understand the nature, risk, meaning, and consequences of the clinical trial (cf. MPG § 20 Sec. 2 Sentence 1 No. 1)
* Chronic kidney disease stage 5D (end stage renal disease) on hemodiafiltration as extracorporeal renal replacement therapy

Study-specific:

* On high volume online (>21 L/session substitution volume postdilution per session) hemodiafiltration (HDF), at least 4 h treatment time thrice weekly ≥3 month
* Vascular access (fistula or graft) and high flow double lumen catheter which enables suitable effective blood flow rate (≥ 300 ml/min)

Exclusion Criteria:

General:

* Any condition which could interfere with the patient's ability to comply with the study. This decision is at the discretion of the treating physician and relates to the general stable condition of the patient (e.g. any acute condition, e.g. infection or mental problem which might give reason for concern etc.)
* Ongoing participation in an interventional clinical study during the preceding 30 days
* Previous participation in this study
* Pregnancy or lactation period
* Patient is not able to give informed consent according to MPG § 20 Sec. 2 Sentence 1 No. 1

Study-specific:

* Recurrent episodes of vascular access failure characterized by e.g. repeated cannulation problems or unstable blood flows within the last 2 months prior to study start (>3 times, respectively)
* Single needle treatments
* Catheter as vascular access (except high flow double lumen catheter)
* Unstable patients (due to e.g. acute intercurrent disease like myocardial infarction, cerebrovascular accident, peripheral arterial occlusion, active malignant disease, use of antibiotics within the last 4 weeks)
* Patients with heart failure (NYHA ≥ 3), COPD (GOLD 2-4), frequent intradialytic symptomatic hypotension requiring intervention within the last 2 months prior to study start (>3 times, respectively)
* Patients with known or suspected allergy to trial product and related products
* Patients with chronic antiallergic medication due to immune-mediated disease
* Planned absence from dialysis unit within the 4 weeks of study duration e.g. due to scheduled hospitalization, holidays or any other reason
* Active HBV, HCV, HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Removal rate of β2-microglobulin | t=240 minutes of HDF
  Removal rate of β2-microglobulin in Plasma related to the albumin removal into the dialysate

CONTACTS AND LOCATIONS:
Overall Officials: Götz Ehlerding, Dr med, Principal Investigator — Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen
Locations (4):
- Germany (4):
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - PHV-Dialysezentrum Goslar, Goslar
  - Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen, Hanover
  - PHV Dialysezentrum Kiel, Kiel